CLINICAL TRIAL: NCT04587700
Title: Analgesic Consumption in Chronic Marijuana Users Following Orthopedic Trauma Surgery
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00102596
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Cannabis; Marijuana
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-marijuana user: Has never consumed marijuana or has abstained for at least the past 12 months
- Chronic Marijuana User: Has used marijuana in any form at least once a week for the past 3 months

SUMMARY:
Marijuana use has increased since its legalization in Canada and many believe that it may help patients that are experiencing chronic pain. The investigators want to assess if patients who have used marijuana chronically will need more medication to control their pain after they have undergone orthopedic trauma surgery (ex. Hip, femur, humerus fractures etc.). In this study, the investigators will identify chronic marijuana users (ie. those using for 3 months or more) who are undergoing orthopedic trauma surgery to assess how much pain medication they need post-operatively and compare this with non-users. The investigators will also evaluate their pain scores, pain medication use and other complications that they may have during or after their surgeries, including any nausea/vomiting, heart or breathing problems.

DETAILED DESCRIPTION:
Since its legalization in Canada, marijuana consumption has become more common while also being the most widely used illicit drug within the USA. In addition to being consumed recreationally, cannabis is being increasingly prescribed by medical practitioners as nearly 15% of Canadian and Australian patients experiencing chronic pain use it as one component of treatment. Recent evidence has demonstrated that specific patient cohorts may benefit from cannabis, including those with fibromyalgia, diabetic neuropathy, complex regional pain syndrome, multiple sclerosis, traumatic neuropathic pain, and difficulty sleeping due to chronic pain, amongst others. Cannabis contains two main components: delta-9-tetrahydrocannabinol (THC), which is active, and cannabidiol, which is inactive. THC has its effects by binding to Type 1 cannabinoid receptors and inhibiting pain pathways while activation of Type 2 cannabinoid receptors have anti-inflammatory properties.

As literature continues to investigate its analgesic characteristics, many proponents of cannabis use believe that it can modify pain response in various settings. One such setting that is of special interest for pain control is during the post-operative period. Currently, there is minimal data available to reflect the analgesic requirement, and thus degree of pain, for a patient who is a chronic marijuana user immediately following a surgical procedure. A class of surgical procedures that is of particular interest to us due to its pain-evoking characteristics is orthopedic trauma surgery. In fact, orthopedic surgeons are one of the higher opioid prescribing specialists, potentially highlighting the difficulty in achieving adequate pain control in their patient population. More information is required to better tailor analgesia for these patients as it may contribute towards their overall recovery, restoring mobility, and patient satisfaction (6,7).

Through this study, the investigators would like to investigate the relationship between orthopedic trauma surgery and post-operative pain control in the chronic marijuana user. Minimal data is available in the literature reflecting this potentially common situation. Specifically, the investigators are interested in the clinical implications of marijuana use on opioid consumption and verbal pain rating in this patient scenario. The investigators also hope that the data can reflect possible side effects or other concerning outcomes in the peri-operative period so that clinicians may be able to provide more personalized care to these patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults ranging from age 18-75 years old
* Patients undergoing orthopedic trauma surgery
* Patients who consent to the study
* ASA class I to III

Exclusion Criteria:

* Patient refusal
* Patients lacking capacity to consent
* Intraoperative regional anesthesia technique
* Chronic pain patient

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient recruits will be identified by accessing the electronic health record at the University of Alberta hospital (Edmonton, Alberta, Canada) and the written slate available at the Royal Alexandra hospital (Edmonton, Alberta, Canada). These sources will list the elective orthopedic slate, accessible about 1 week prior to surgery, and the trauma slate which is available at least 24 hours prior to surgery. Patients can also be identified in the pre-assessment clinic. Research supervisors and designated assistants will be responsible for identifying potential participants. Once their location is identified, the research assistant will consent the patient at least 12 hours prior to surgery or in the pre-assessment clinic where patients will attend at least 24 hours prior to surgery.
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-07-05 (Actual)

PRIMARY OUTCOMES:
Total opioid consumption | Within 24 hours post-operatively
  The total opioid consumption (morphine equivalents) at 24 hours post-operatively in chronic marijuana users compared to the control group (no marijuana).

CONTACTS AND LOCATIONS:
Overall Officials: Vivian Ip, MBChB, Principal Investigator — Staff Anesthesiologist
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada